CLINICAL TRIAL: NCT01582620
Title: Telestroke in Nordland Hospital: Improved Treatment of Cerebral Stroke in Small Hospitals
Brief Title: Telestroke in Nordland Hospital. A Study of a Telemedicine Network in Rural Hospitals
Acronym: Telestroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator moved, and the study should have been taken out of UNN Clincaltrial.gov account 5-6 years back in time.
Sponsor: University Hospital of North Norway (Other)
Collaborators: Nordlandssykehuset HF (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010/2277(REK); 2277/2010 (REK) (Other: The National Committees for research ethics in Norway)
Record Dates: First submitted 2011-05-26; First posted 2012-04-20 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2012-04

CONDITIONS: Stroke, Acute
Keywords: Cerebrovascular disorders; Telemedicine; remote consultation; rural; thrombolysis therapy; plasminogen activators; stroke care; stroke management
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Telestroke — remote videoconference consultations

SUMMARY:
The purpose is to study the clinical, technological and organizational impacts of a telestroke service between Nordlandssykehuset, Bodø, and two small rural hospitals in Lofoten and Vesterålen. The stroke specialist in Bodø will examine the patient in cooperation with the doctor at the local hospital through video- and sound communication. Radiology images are transmitted using the RIS/PACS system.

Telestroke consultations may be useful to assess whether the patient needs thrombolysis medication, and also whether there is a need for more advanced specialist neurological or neurosurgical treatment, supporting quick triaging and transfer to the appropriate unit.

The study design is a multi-method approach using before-and-after hospital information data as well as registration forms monitoring patient outcome and pathways. The research questions will be approached from medical, organisational and technological perspectives.

A telestroke service in North Norway is expected to face other challenges than those reported internationally: In Nordlandssykehuset, as in Helse Nord in general, the number of cases is low, clinicians have high turnover, technical support is not available 24/7 and severe weather conditions and long distances might add to the transport time.

Primary hypothesis: The use of telestroke leads to faster and more accurate diagnosis and proper treatment

Secondary hypothesis: Telestroke leads to improved overall patient treatment

DETAILED DESCRIPTION:
There is good evidence that the prognosis for patients with ischemic stroke is improved by thrombolysis in the acute phase. The challenge is the narrow time window: Thrombolysis should be given as soon as possible and not later than 4.5 hours after the first symptoms. In Norway, only approximately 2% of all stroke patients receive thrombolysis whereas 20 % are expected to benefit from such treatment (The Norwegian Directorate of Health, 2010). The low rate could be due to geographical conditions with long travel distances, lack of awareness in the population, but also little experience with the treatment in local hospitals may play a role.

The overall aim of this project is to improve health outcome for stroke patients by telemedicine. This study will investigate the potential outcome for stroke patients in small rural hospitals using a telestroke service.

The project will study the "patient flow" by analysing hospital information system (HIS) data as well as monitoring the teleconsultations and logging the main purpose for and results of the consultation. This will be conducted throughout the project, and analysed for a period of 18 months. Hospital data on diagnosis, thrombolysis frequencies, stroke complications like haemorrhage or stroke recidive, will be used in the analysis process.

Around 60 cases may potentially be included in the study during the 18 month observation period, which can be compared with register data from patients before the study. Control-groups have been considered, but found not ethical since the telestroke equipment is already installed in the two hospitals.

Log information from the Norwegian Health Net on the use of videoconferencing will be used as a basis for field observations and interviews and to verify the actual use of the system.

Corresponding with the logged data, semi-structured interviews will be conducted by making follow-up phone calls to hospital staff after the telestroke incidents. Using a qualitative approach, the number of follow-up calls will be decided in the process, adding up to app 20 cases. This method will be used to capture what happened in the concrete telestroke incident from the first call to the hospital and throughout the process, while the details of the session are still fresh. There will also be periods of fieldwork at all three hospitals. This will include observations at the hospital wards and during concrete telestroke consultations. Semi-structured focus groups interviews will be conducted with health personnel involved with stroke-patients, including ambulance personnel, doctors and nurses, as well as technical support. Fieldwork will take place early in the project phase, and then at intervals during the project period. Fieldwork and follow-up phone interviews at different times in the research period will capture potential changes in the stroke treatment over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the two local hospitals diagnosed with acute cerebral stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of stroke patients receiving thrombolysis treatment after the introduction of a telestroke service | Approx. 30 months

SECONDARY OUTCOMES:
Door-to-(thrombolysis)needle-time | 18 months
Scores for functional outcomes at admission and discharge | 18 months
Proportion of patient transfers from Lofoten and Vesterålen in the acute phase to secondary level | 18 months
Proportion of stroke patients receiving "telestroke" examination | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Jacobsen, Study Director — Norwegian center for integrated care and telemedicine, Tromsø Norway; Rolf Salvesen, PhD professor, Principal Investigator — Neurological department, Nordlandssykehuset HF; Stein Roald Bolle, PhD, Study Chair — Norwegian center for integrated care and telemedicine, University Hospital North Norway, Tromsø
Locations (2):
- Norway (2):
  - Nordlandssykehuset HF Lofoten, Gravdal, Nordland
  - Nordlandssykehuset HF Vesterålen, Stokmarknes